CLINICAL TRIAL: NCT07048197
Title: An Open-label, Multi-center, Phase 1/2 Study to Assess Safety, Cellular Kinetics and Exploratory Efficacy of Rapcabtagene Autoleucel in Participants With Difficult-to-treat Rheumatoid Arthritis and Severe, Refractory Sjogren's Disease With Organ Involvement
Brief Title: A Study to Assess Safety, Cellular Kinetics and Exploratory Efficacy of Rapcabtagene Autoleucel in Rheumatoid Arthritis and Sjogren's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323M12101B; 2024-514596-18-00 (Other: EU CT)
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA) and Sjögren's Disease (SjD)
Keywords: CAR-T,; YTB323,; rapcabtagene autoleucel,; D2T RA,; srSjD
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapcabtagene autoleucel-rheumatoid arthritis (Experimental): Single infusion of Rapcabtagene autoleucel in participants with rheumatoid arthritis
  Interventions: Biological: Rapcabtagene autoleucel
- Rapcabtagene autoleucel- Sjögren's Disease (Experimental): Single infusion of Rapcabtagene autoleucel in participants with Sjögren's Disease
  Interventions: Biological: Rapcabtagene autoleucel

INTERVENTIONS:
Biological: Rapcabtagene autoleucel — Single infusion of Rapcabtagene autoleucel

SUMMARY:
A study to assess safety, cellular kinetics and exploratory efficacy of rapcabtagene autoleucel in rheumatoid arthritis and Sjogren's disease

DETAILED DESCRIPTION:
The study is intended to assess safety, cellular kinetics and any early sign for efficacy of rapcabtagene autoleucel in participants with difficult-to-treat rheumatoid arthritis (D2T RA) and severe, refractory Sjogren's disease (srSjD) with organ involvement.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Men and women aged ≥ 18 years and ≤ 75 years at Screening For RA only
* Diagnosis of rheumatoid arthritis
* Treatment failure of standard of care therapies
* Active disease For SjD only
* Diagnosis of Sjogren's disease
* Active disease

Exclusion Criteria:

* BMI at Screening of ≤17 or ≥ 40 kg/m2
* Clinically significant active, opportunistic, chronic or recurrent infection
* Sexually active males unwilling to use a condom during intercourse from the time enrollment
* Women of childbearing potential, unless they are using a highly effective method of contraception starting from the time of enrollment
* Female participants who are pregnant, breastfeeding or intending to conceive during the course of the study
* Inadequate organ function during screening
* History of lymphoproliferative disease or any known malignancy or history of malignancy
* History of bone marrow/hematopoietic stem cell or solid organ transplantation
* Any psychiatric condition or disability making compliance with treatment or informed consent impossible

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 months
  Safety parameters include vital signs, adverse events, laboratory parameters and ECG evaluation

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter: Cmax | 24 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Maximum observed blood concentration Cmax).
PK parameter: Tmax | 24 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Time to reach maximum concentration Tmax).
PK parameter: T1/2 | 24 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Terminal elimination half-life T1/2).
PK parameter: Clast | 24 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Last measurable concentration Clast).
PK parameter: Tlast | 24 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Time to reach last measurable concentration Tlast).
PK parameter: AUC | 24 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Area under plasma concentration -time AUC).

CONTACTS AND LOCATIONS:
Locations (10):
- France (4):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid